CLINICAL TRIAL: NCT04985474
Title: Impact of Pulmonary Rehabilitation After Lung Resection for Cancer on Patients' Level of Anxiety and Depression
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 15-METHODO-02
Record Dates: First submitted 2016-09-13; First posted 2021-08-02 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Pulmonary Resection
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pulmonary resection
  Interventions: Other: questionnaires

INTERVENTIONS:
Other: questionnaires

SUMMARY:
The interest of pulmonary rehabilitation for patients who underwent lung resection for cancer remains controversial. The investigators studied the effects of the RR and its impact on quality of life and level of anxiety and depression in patients.

In 2011 and 2012 , an RR was proposed to the patients referred to our center after lung resection for cancer. Patients were assessed at entry and departure by 6minutes walk test , a visual analog pain scale , a quality of life questionnaire ( EORTC QLQ C30 ) and an anxiety questionnaire and Depression (HAD) . These same questionnaires were mailed 6 months after the end of the pulmonary rehabilitation .

ELIGIBILITY:
Inclusion Criteria:

* Patient with pulmonary resection
* Patients undergoing a standardized approach (or thoratomie videothoracoscopy)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing a standardized approach (or thoratomie videothoracoscopy)
Sampling Method: Non-Probability Sample
Enrollment: 133 (Actual)
Dates: Start 2011-01; Primary Completion 2011-01 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
level of depression with scale | At 6 months
  Assess the level of depression during and after a respiratory rehabilitation training in institutions
level of anxiety withe scale | At 6 months
  Assess the level of anxiety during and after a respiratory rehabilitation training in institutions